CLINICAL TRIAL: NCT07127562
Title: Effect of a Simplified Mindfulness Intervention on Health-related Quality of Life in Patients Undergoing Hematopoietic Stem Cell Transplantation: A Prospective Single-Center Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2025078
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness intervention group (Experimental): 1. Mindfulness intervention group: Intermittent period: from the first day to at least the 21st day, and up to the 28th day, continuous implementation
  Content of intervention (daily completion):
  1. Mindfulness breathing exercise (10 minutes) Content: Close your eyes to perceive the breath coming in and out, pay attention to the present moment, without judgment; Tools: Chinese voice-guided audio (nurses check room or patients scan code to play); Time: to be completed between 9am and 10am;
  2. Body Scan Exercise (15 minutes) Content: gradually perceive the tension, pain or relaxation of each part of the body from head to toe; Tools: Chinese audio guidance, which can be played during the infusion or before going to bed; Time: between 7-8pm;
  Interventions: Behavioral: Mindfulness intervention
- Conventional support group (No Intervention): received conventional nursing and rehabilitation guidance, but did not receive mindfulness intervention. The control group patients received conventional hospital nursing services during the study period, including disease monitoring, drug treatment, rehabilitation guidance, etc., but did not receive any form of mindfulness training or other similar psychological interventions.

INTERVENTIONS:
Behavioral: Mindfulness intervention — Intermittent period: from the first day to at least the 21st day, and up to the 28th day, continuous implementation
  Content of intervention (daily completion):
  1. Mindfulness breathing exercise (10 minutes) Content: Close your eyes to perceive the breath coming in and out, pay attention to the present moment, without judgment; Tools: Chinese voice-guided audio (nurses check room or patients scan code to play); Time: to be completed between 9am and 10am;
  2. Body Scan Exercise (15 minutes) Content: gradually perceive the tension, pain or relaxation of each part of the body from head to toe; Tools: Chinese audio guidance, which can be played during the infusion or before going to bed; Time: between 7-8pm;
  Arms: Mindfulness intervention group

SUMMARY:
This study aims to evaluate the impact of a simplified mindfulness intervention (daily mindfulness breathing and body scanning) during hospitalization in the transplant ward on health-related quality of life in hematopoietic stem cell transplantation patients.

DETAILED DESCRIPTION:
All patients undergo standardized HSCT treatment, which does not interfere with the management of their underlying conditions. Patients are randomly assigned to either the 'Mindfulness Intervention Group' or the 'Conventional Support Group' based on age (whether over 40) and transplant type (autologous or allogeneic), in a 1:1 ratio. The study period is at least 21 days, during which patients are hospitalized in the transplant ward.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Scheduled to receive either autologous or allogeneic HSCT.
3. Anticipated inpatient stay in the transplant unit of at least 21 days.

Exclusion Criteria:

1. Prior history of hematopoietic stem cell transplantation (HSCT).
2. Active psychiatric disorder or cognitive impairment.
3. Systematic training in mindfulness/mindfulness-based interventions/yoga within the past 3 months.
4. Contraindications to MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-08-07 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in FACT-BMT Score (Δ Score) | baseline to Day 28
  The daily trajectory of FACT-BMT total scores during hospitalization will be continuously monitored in both the mindfulness intervention group and the routine support group. The difference between the lowest daily score and the baseline score (Δ nadir) will be calculated to reflect the maximum decline in quality of life during hospitalization. A comparison will be made between the two groups to determine whether there is a difference in the maximum reduction of FACT-BMT total scores during hospitalization, thereby evaluating the mitigating effect of mindfulness intervention on the deterioration of quality of life.

SECONDARY OUTCOMES:
Change in HADS score | Baseline, Day 28
  Assessing trends in emotional improvement.
EQ-5D-5L score | baseline ，Day 28
  Includes 5-dimensional scores and Visual Analog Scale (VAS) ratings to reflect subjective health status
MoCA cognitive function | baseline ，Day 28
  Evaluating cognitive performance.
MRI structural changes | Day 0, Day 28
  Hippocampal volume, dorsolateral prefrontal cortex (DLPFC) thickness, and surface area
Incidence of bloodstream bacterial infections in the transplant unit | From Day 0 through discharge
  Including the number of positive bacterial blood cultures
Post-Traumatic Growth Inventory (PTGI) | baseline, Day 28
  Assessing the degree of personal growth following traumatic experiences
Subjective Well-Being Scale (SWB) | baseline, Day 28
  Measuring life satisfaction and quantifying emotional experiences
Pittsburgh Sleep Quality Index (PSQI) | baseline, Day 28
  Quantifying sleep quality